CLINICAL TRIAL: NCT05983692
Title: Clinical Translation of Biodegradable Magnesium Wire for Augmentation of Anterior Cruciate Ligament (ACL) Reconstruction From Bench Side to Bedside: A Multicentre, Double-blinded, Randomised Controlled Trial
Brief Title: Mg Wire for Augmentation of ACL Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Alice Ho Miu Ling Nethersole Hospital (Other); Kwong Wah Hospital (Other); Tseung Kwan O Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021.654
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACLR; Mg wire; Bone tendon interface healing
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mg Wire group (Experimental): Intervention: Magnesium-based wire as braiding suture to braid the tendon graft.
  Interventions: Device: Magnesium based wire
- control group (No Intervention): 2-0 vicryl suture as control, size and length matched Mg wire

INTERVENTIONS:
Device: Magnesium based wire — Mg wire will be used as a braiding suture to braid tendon graft, which is a standard preparation of graft and is not related to fixation of the tendon graft
  Arms: Mg Wire group

SUMMARY:
Background: ACLR with autologous tendon graft is commonly used for the treatment of ACL injury. However, as the BTI healing is poor, this can lead to a failure rate of 5% in the first-year post-operation; a long and unpredictable rehabilitation period is expected and 35 % of patients never return to preinjury level of sports. Biological enhancement of BTI healing will help to cut down the medical cost related to poor prognosis. As a biodegradable metal, Mg has been developed as implants in orthopaedics for decades, yet without clinical implants developed for ACLR. Our team has been working on this area in the past 10 years preclinically. Our animal studies showed that supplementation of magnesium wire significantly promotes osteogenesis at BTI and improves mechanical strength in ACLR. Recently, our team developed a highly pure (99.99%) Mg wire (Fig 2) in collaboration with metallic engineers for tendon graft braiding during ACLR and with its improved physical quality and strength, it is suitable for graft braiding and then its degradation in vivo can promote tunnel bone formation and bone tendon interface integration.

Objective: To investigate if anterior cruciate ligament (ACL) reconstruction augmented with magnesium (Mg) wire enhances osteogenesis at the bone-tendon interface (BTI), improving post-op rehabilitation and leading to better clinical outcomes.

Hypothesis: Patients with ACL reconstruction using Mg wire will experience improved osteogenesis at the BTI, more effective rehabilitation, and superior knee strength and function.

Design and Subjects: A multicentre, double-blinded, randomized controlled trial will recruit patients aged 18-30 with unilateral ACL tear for primary ACLR with a hamstring graft at four sites.

Instruments: Mg-based wire.

Interventions: Participants will receive either 99.99% purity Mg wire or 2-0 vicryl as a control.

Main Outcomes: Osteogenesis will be assessed by High-Resolution Peripheral Quantitative Computed Tomography (HR-pQCT), muscle strength via Biodex tests, and functional recovery with International Knee Documentation Committee (IKDC) and Tegner scores at multiple post-op intervals. Knee stability will be checked with KT-1000 arthrometer. Blood samples will be analyzed for inflammatory markers and metabolic effects related to Mg wire.

Data Analysis and Expected Results: A repeated-measures ANOVA will be utilized for data analysis. The expectation is that Mg wire augmentation will significantly enhance osteogenesis at the BTI and improve rehabilitation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* Unilateral ACL tear for primary ACLR (Single bundle, Hamstring) confirmed clinically and radiologically.

Exclusion Criteria:

* Concomitant multiple ligament injuries requiring additional surgical procedures,
* Preoperative radiographic signs of arthritis,
* Revision ACLR
* Femoral tunnel interference screws
* Contralateral knee with ACL deficiency or reconstruction
* Medical co-morbidities
* Long-term steroid intake
* Non-compliance to our rehabilitation protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Bone shell size | 2 weeks and 3, 6, 12 and 24 months post-operation.
  HR-pQCT (ExtremCT II, Scanco, Switzerland) will be used to measure the bone shell size at graft tunnel interface. The involved knees will be investigated. A total of 1344 axial slices with an image matrix of 2304 × 2304 were collected at a nominal isotropic voxel size of 60.7μm. The scan region was defined by the scout view image acquired in the sagittal plane.The total scanning length was 81.6mm which covered the tunnel from proximal tibia to distal femoral condyle (X-ray settings: 68kVp, 1470μA, 100ms integration time, 156mAs per stack (168 slices).Image segmentation will be performed to select the bone shell features at graft tunnel interfaces near femoral and tibial intra-articular apertures with standardized threshold values at a thickness of ~2.5 mm (40 slices). Geometric transformation will be performed to adjust for the variations in angle between scanning axis and tunnel axis by a cosine function.

SECONDARY OUTCOMES:
International Knee Documentation Committee | Pre-operation, 2 weeks and 3, 6, 12 and 24 months post-operation.
  Consists of 10 questions on symptoms and activity ranging from 0 to 100 where 100 implies perfect knee function.
Tegner activity score | Pre-operation, 2 weeks and 3, 6, 12 and 24 months post-operation.
  This is an activity level scaled from 1 (low activity) to 10 (high activity).
Passive Knee laxity | 3, 6, 12 and 24 months post-operation.
  To measure anterior-posterior knee laxity, the KT-1000 knee ligament arthrometer (MEDmetric Corp, San Diego, CA, USA) will be used. A manual force test will be applied until a 30lb sound signal is activated. Three trials will be performed. A side difference of 3 mm above is considered clinically relevant.
Isokinetic muscle strength | 3, 6, 12 and 24 months post-operation
  The dynamometer (Biodex System 4, Biodex Medical Systems Inc., New York, USA) will be used for measuring Isokinetic muscle strength in N. Subjects will perform a standardized warm-up exercise (5 min cycling) followed by the test. Concentric/concentric contractions of knee extension/flexion will be tested at 60°/s and 180°/s. Subjects will be seated on the dynamometer chair with their hips flexed to 85°.
Cytokines assay | Pre-operation, Day 1, 2 and 6 weeks and 3 months post-operation
  To evaluate the safety of Mg wire with respect to inflammatory responses, 5 ml blood samples will be collected for C-reactive protein measurement using ELISA kit.
  Measurements of Ca, Mg, P, Cr, Urea, ALT, AST, TP, ALB, GLB will be taken to monitorpotential effect of the Mg wire. The blood tests will be performed at baseline, day 1 post-op, 2 weeks, 6 weeks and 12 weeks post-op, since the degradation of Mg wire is faster based on our preclinical study results.
Single leg hop distance | 6, 12 and 24 months post-operation
  The average of single leg hop distance in cm with three attempts will be measured during the single leg hop test.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers